CLINICAL TRIAL: NCT02218476
Title: Beneficial Effects of Coenzyme Q10 Treatment on the Mitochondrial Dysfunction and Oxidative Stress Associated to Atherothrombosis Developement in Antiphospholipidid Syndrome Patients
Acronym: coenzyme Q10
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Maimónides Biomedical Research Institute of Córdoba (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: PI12-01511
Record Dates: First submitted 2014-08-08; First posted 2014-08-18 (Estimated); Last update posted 2014-08-18 (Estimated); Status verified 2014-08

CONDITIONS: Coenzyme Q10 on Athero-thrombosis in APS Patients
MeSH Terms: interventions — coenzyme Q10

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (1):
- APS Patient (Other)
  Interventions: Drug: CoQ10; Drug: Placebo

INTERVENTIONS:
Drug: CoQ10
Drug: Placebo

SUMMARY:
The study will be performed on 50 APS (antiphospholipid Syndrome) patients, which will be randomized to receive either CoQ10 (200mg/day) or placebo for one month. Blood will be drawn at time 0 and at the end of the treatment. Studies will be conducted in plasma and purified leukocytes from APS. Design: 1) Study of endothelial function: 2) Analysis of changes operated on various prothrombotic/proinflammatory parameters and their associated intracellular signalling. 3) Analysis of mitochondrial ultra structure and activity; mitochondrial antioxidant system characterization; Expression levels and activity of transcription factors/proteins involved in oxidative stress (Foxo 3, NFkB, Nrf2), Quantification of CoQ10 (Coenzyme Q10). 4) Biomarkers of oxidative stress. 5) miRNAs microarrays, RT-PCR validation and correlation/association studies. 6) Induction of over-expression of miRNAs of interest; luciferase constructs. 7)Studies of methylation.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who fulfilled Sidney criteria for APS (antiphospholipid Syndrome) (Miyakis S et al., J Thromb Haemost 2006; 4:295-306)
2. Age over 18 years
3. Written informed consent

Exclusion Criteria:

1. Acute Liver Disease.
2. Severe renal impairment
3. Acute arterial or venous thrombosis episode in the last 3 months
4. Pregnancy and breastfeeding

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50
Dates: Start 2013-09; Primary Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
Change in endothelial function in vivo | 0 weeks, 4 weeks, 8weeks, 12weeks
  Study of the endothelial function in vivo. Variations in capilar blood flow of the skin will be analyzed by noninvasive Doppler laser fluorimetry using a Periflux 5000 equipment.
  The study will be performed on 50 APS (antiphospholipid Syndrome) patients. Patients will be randomized to CoQ10 or placebo group. Treatments will be given for 1 month, according to a randomized and crossover design (with wash-out periods of four weeks) Blood will be drawn at time 0, at the end of treatment, and after three months of the end of treatment.

SECONDARY OUTCOMES:
Change in Tissue factor | 0 weeks, 4 weeks, 8 weeks, 12 weeks
  Parameters related to inflammation and thrombosis in cells measure at mRNA and VEGF (Vascular Endothelial Growth Factor) in serum/plasma and cells.
  The study will be performed on 50 APS (antiphospholipid Syndrome) patients. Patients will be randomized to CoQ10 or placebo group. Treatments will be given for 1 month, according to a randomized and crossover design (with wash-out periods of four weeks) Blood will be drawn at time 0, at the end of treatment, and after three months of the end of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Rosario Lopez Pedrera, Biology, Principal Investigator
Locations (1):
- Hospital Universitario Reina Sofía de Córdoba, Córdoba, Andalusia, Spain

REFERENCES:
- [Derived] Perez-Sanchez C, Aguirre MA, Ruiz-Limon P, Abalos-Aguilera MC, Jimenez-Gomez Y, Arias-de la Rosa I, Rodriguez-Ariza A, Fernandez-Del Rio L, Gonzalez-Reyes JA, Segui P, Collantes-Estevez E, Barbarroja N, Velasco F, Sciascia S, Cecchi I, Cuadrado MJ, Villalba JM, Lopez-Pedrera C. Ubiquinol Effects on Antiphospholipid Syndrome Prothrombotic Profile: A Randomized, Placebo-Controlled Trial. Arterioscler Thromb Vasc Biol. 2017 Oct;37(10):1923-1932. doi: 10.1161/ATVBAHA.117.309225. Epub 2017 Jul 6. PMID 28684614